CLINICAL TRIAL: NCT02532790
Title: The Research of Standard Diagnosis and Treatment for Henoch-Schonlein Purpura Nephritis With Mild Proteinuria in Children
Brief Title: The Research of Standard Diagnosis and Treatment for HSPN With Mild Proteinuria in Children
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Nanjing Children's Hospital (Other)
Responsible Party: Principal Investigator, Aihua Zhang, Hospital vice president, Nanjing Children's Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: AiZhang
Record Dates: First submitted 2015-08-20; First posted 2015-08-26 (Estimated); Last update posted 2020-02-26 (Actual); Status verified 2020-02

CONDITIONS: Henoch-Schoenlein Purpura Nephritis
Keywords: Mild proteinuria
MeSH Terms: interventions — Prednisone; benazepril

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- group 1 (Experimental): Prednisone Drug : prednisone 1.5mg/kg/d for 4-6 weeks, then 1.5mg/kg/d qod for 4 weeks, reduce 5mg every 2-4 weeks If the proteinuria decreases by less than 50% after treating for two months, this candidate reaches the ending point.
  Interventions: Drug: Prednisone
- group 2 (Experimental): Angiotension converting enzyme inhibitors(ACEI) Drug: lotensin 0.2-0.3mg/kg/d (the maximum dose is 20mg)
  Interventions: Drug: ACEI

INTERVENTIONS:
Drug: Prednisone — 1.5mg/kg/d
  Arms: group 1
Drug: ACEI — 0.2-0.3mg/kg/d
  Other Names: Lotensin
  Arms: group 2

SUMMARY:
This study is performed to evaluate the efficacy and safety of various measures in the treatment of HSPN with mild proteinuria in children.

DETAILED DESCRIPTION:
Henoch-Schonlein purpura nephritis (HSPN) is one of the most common complications of Henoch-Schonlein purpura, and has become one of the main causes of chronic kidney disease in children. However, the diagnosis and treatment of HSPN is still based on the clinical experience, lacking of evidence-based support. This study is performed to explore the biological markers for early prediction of the prognosis and evaluate the efficacy and safety of various measures in the treatment of HSPN in children.

The patients who are proved to get HSPN by renal biopsy will be randomized to receive either prednisone p.o. or angiotensin-converting enzyme inhibitor(ACEI) p.o. We will follow up them for about 2.5 years and compare the efficacy and safety of both measures by monitoring several indexes.

ELIGIBILITY:
Inclusion Criteria:

* Renal biopsy proved HSPN (ISKDC class II)
* Proteinuria < 25 mg/kg/d

Exclusion Criteria:

* The children with congenital diseases
* Proteinuria≥25 mg/kg/d

Ages: 2 Years to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 100 (Estimated)
Dates: Start 2015-08; Primary Completion 2020-07 (Estimated); Study Completion 2020-07 (Estimated)

PRIMARY OUTCOMES:
Disappearance of proteinuria | 30 months
  The proteinuria is < 150mg/d

SECONDARY OUTCOMES:
Disappearance of hematuria | 30 months
  The number of red blood cells is < 3 in each high power field of vision
Renal function | 30 months
  The glomerular filtration rate is normal

CONTACTS AND LOCATIONS:
Overall Officials: Aihua Zhang, M.D., Study Chair — Department of Nephrology, Nanjing children's hospital
Locations (1):
- Nanjing Children's Hospital, Nanjing, Jiangsu, China

REFERENCES:
- [Derived] Hahn D, Hodson EM, Craig JC. Interventions for preventing and treating kidney disease in IgA vasculitis. Cochrane Database Syst Rev. 2023 Feb 28;2(2):CD005128. doi: 10.1002/14651858.CD005128.pub4. PMID 36853224